CLINICAL TRIAL: NCT01245244
Title: Morphine Modulation of The Brain's Pain Matrix
Acronym: Mor2010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2010-020894-17
Record Dates: First submitted 2010-09-24; First posted 2010-11-22 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Experimental)
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator)
  Interventions: Other: orange juice

INTERVENTIONS:
Drug: Morphine — Morphine oral mixture
  Other Names: Morphine hydrochloride oral solution 2 mg/ml
  Arms: Morphine
Other: orange juice — orange juice
  Other Names: orange juice solution
  Arms: Placebo

SUMMARY:
The aim of the current project is to use a model of painful stimulation of skin, muscles and internal organs, where it is possible to measure activity in the brain centers that process pain simultaneously. Magnetic resonance imaging and electroencephalography are combined to optimize the anatomical and physiological description of brain activation. During administration of morphine we will identify how different brain areas are affected. This knowledge will be used to:

1. Understand the mechanisms of morphine to a greater extent than is possible today, including:

1. to investigate the mechanisms of morphine versus placebo on pain signals in the spinal cord and brain. This is done by a combination of experimental pain models, neurophysiological and imaging techniques (EEG and fMRI). This can be achieved as both subjective and objective measures of the analgesic effect.
2. to examine morphines effect on communication between the centers of the brain that are involved in painprocessing .
3. modeling of morphine pharmacokinetics (the understanding of what the body does to the drug, such as. concentration in the blood and the brain), since this is central to understand the pharmacodynamics (the description of what the drug does to the body and thus the effect it has).
4. to identify biomarkers that can predict whether healthy subjects respond to morphine by experiencing an analgesic effect.

DETAILED DESCRIPTION:
The tests will consist of one main study (I) and one sub-study (i):

I) Experiments in the painlaboratory in the gastroenterology clinic, where 40 healthy subjects will be examined with different pain tests i) Experiments in the MRI scanner, where only 20 of the 40 from the main study will be investigated in a more simple pain model. The individuals who also participate in MRI studies, will consist of those who first sign up

An equal distribution of men and women is wanted. The trial will be a double-blind, placebo-controlled crossover study in which all subjects will be investigated on two seperate days and receive respectively placebo or morphine in random order

Skin stimulation

Skin will be stimulated with thermal and electrical stimuli. Stimulated by:

* Thermal stimuli by the skin stimulated with heat with an approved termotester (Medoc termotest) or with cold, by a hand or foot immersed in ice water. This harmless ice water test is further possible to evaluate DNIC (diffuse noxious Inhibitory controls) which is part of the pain system descending inhibitory system.
* Electrical stimulation of the skin will be done by: 1) to the skin of the forearm stimulated electrically through two small surface electrodes (each approx. One cm2). There are stimulated to pain threshold, 2) via surface electrodes placed under the foot. This activates the nociceptive avert reflex as recorded by electrodes placed on the leg.

Muscle stimulation

The muscles can be stimulated by:

• mechanical stimuli by pressing the muscle with an approved pressure algometer (Somedic produktion AB, Sweden). There is an upper limit for the pressure to avoid injury.

Bone stimulation

Bone associated pain can be studied by:

• mechanical stimuli by pressing the right shin bone 15cm below the patella, medial of the tibia. Pressed with a handheld trykalgometer (Type 2, Somedic produktion AB, Sweden) with a probe size of 2mm in diameter until trial participants reach their pain tolerance threshold.

Visceral stimuli Stimuli to the rectum will be performed through the probe specifically designed for this purpose.

* mechanical stimuli will be applied by water filling a balloon which is glued on the probe. The balloon on the probe is extended to moderate pain. The expansion is done by slowly filling the balloon with 37 degrees hot water.
* Thermal stimuli will be applied by flushing the balloon with hot water (60 ° C)
* Electrical stimuli will be applied by stimulation of the mucosa with weak electrical currents (Less than 80 mA) through electrodes on the probe. This stimulus is also used for recording of evoked brain potentials.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated "Written informed consent"
2. Age between 20 and 65.
3. Caucasian
4. That it is in the researcher's belief that the subject fully understand the contents of the study and is willing and able to comply with instructions, have the opportunity to meet with visitors, and is expected to complete the entire study. Further, it is in the researcher's beliefs (by which demanded strict action to exclusion criterion 4 and 5) that subjects with abusive tendencies are not included .
5. The person must be healthy ie. without previous chronic or recurrent pain rewarding diseases. Including the person must have:

   1. a blood pressure is 140/90 or less. If not satisfied, a medical assessment to determine whether the person is still included, albeit with a comment and reasons recorded in the CRF.
   2. a resting heart rate of at least 45 bpm. minute (measured after 5 minutes of recumbent rest). If not satisfied, a medical assessment to determine whether the person is still included, albeit with a comment and reasons recorded in the CRF.
6. That women use safe contraceptive methods as the pill, coil, depot injection of progestin subdermal implantation, hormonal vaginal ring and transdermal patch.
7. Negative pregnancy test prior to the conclusion of the experiment

Exclusion Criteria:

1. Pregnancy.
2. Known allergy to study medication
3. Current or previous participation in another drug trial within 30 days before screening.
4. Former participation in trials when given morphine or morphine-like substances.
5. Former addiction behaviors defined as abuse of alcohol, marijuana, opiates or other narcotics or family members who have been / are a drug addict.
6. Earlier pain rewarding or mental illness.
7. Expected need for medical treatment, surgery or hospitalization during the study
8. Concomitant use of strong pain medications
9. Use of any analgesics 24 hours before each test.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Morphine modulation of composite pain assessments | october 2010 - december 2012

SECONDARY OUTCOMES:
Side effects of morphine | october 2010 - december 2012

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Olesen, PhD, Study Chair — Aalborg University Hospital
Locations (1):
- Department of Gastroenterology, Aalborg Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Hansen TM, Olesen AE, Graversen C, Drewes AM, Frokjaer JB. The Effect of Oral Morphine on Pain-Related Brain Activation - An Experimental Functional Magnetic Resonance Imaging Study. Basic Clin Pharmacol Toxicol. 2015 Nov;117(5):316-22. doi: 10.1111/bcpt.12415. Epub 2015 May 29. PMID 25924691
- [Derived] Hansen TM, Graversen C, Frokjaer JB, Olesen AE, Valeriani M, Drewes AM. Single-sweep spectral analysis of contact heat evoked potentials: a novel approach to identify altered cortical processing after morphine treatment. Br J Clin Pharmacol. 2015 Jun;79(6):926-36. doi: 10.1111/bcp.12579. PMID 25556985